CLINICAL TRIAL: NCT00919516
Title: Use of Autologous Bone-Marrow Mononuclear Cell Implantation Therapy as a Limb Salvage Procedure in Patients With Moderate to Severe Peripheral Arterial Disease
Brief Title: Autologous Bone Marrow Mononuclear Cell Implantation for Moderate to Severe Peripheral Arterial Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Vascular and Vein Center, Columbus, OH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRANZ-07-0046
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Peripheral Arterial Disease
Keywords: Bone marrow transplantation; Ischemia; Neoangiogenesis; Peripheral arterial disease; Stem cell therapy
MeSH Terms: conditions — Peripheral Arterial Disease; Ischemia; Neovascularization, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell Implantation (Experimental)
  Interventions: Procedure: Bone marrow mononuclear cell implantation

INTERVENTIONS:
Procedure: Bone marrow mononuclear cell implantation — Dual intramuscular and intra-arterial injections of bone marrow mononuclear cells harvested from the iliac crest. Injection sites are determined by location of stenosis and/or occlusion on angiogram obtained prior to implantation and typically occur in three medial and three lateral sites approximating the disease location.

SUMMARY:
The purpose of this study is to evaluate the efficacy of dual intramuscular and intra-arterial autologous bone marrow mononuclear cell implantation for the treatment of patients with moderate to severe peripheral arterial disease in whom amputation was considered the only viable treatment option.

Study Hypothesis: Patients with moderate to severe peripheral arterial disease who receive intramuscular and intra-arterial stem cell injections will have improved ankle brachial index (ABI) measurements; relief of rest pain; ulcer healing, if applicable; and absence of major limb amputations.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Patients with moderate or severe limb-threatening PAD, defined as ankle brachial indices (ABI) less than 0.7 or presence of non-healing ischemic ulcers with stenosis or occlusion of two of the following lower extremity arteries: anterior tibial, posterior tibial, and peroneal.
* Patients with conditions that preclude recommendation of traditional endovascular or open bypass treatments.

Exclusion Criteria:

* Patients younger than 18 years of age.
* Patients who are eligible to undergo traditional endovascular or open bypass for the treatment of PAD.
* Female patients who are or may be pregnant.
* Patients who are prisoners.
* Patients with mental retardation or are unable to consent for participation independently.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-12; Primary Completion 2013-01 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Major limb amputation | three months

SECONDARY OUTCOMES:
Improved ABI measurements | three months
Relief of rest pain | three months
Ulceration healing | three months

CONTACTS AND LOCATIONS:
Overall Officials: Randall W Franz, MD, Principal Investigator — The Vascular and Vein Center
Locations (1):
- The Vascular and Vein Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Franz RW, Parks A, Shah KJ, Hankins T, Hartman JF, Wright ML. Use of autologous bone marrow mononuclear cell implantation therapy as a limb salvage procedure in patients with severe peripheral arterial disease. J Vasc Surg. 2009 Dec;50(6):1378-90. doi: 10.1016/j.jvs.2009.07.113. Epub 2009 Oct 17. PMID 19837539
- [Derived] Franz RW, Shah KJ, Pin RH, Hankins T, Hartman JF, Wright ML. Autologous bone marrow mononuclear cell implantation therapy is an effective limb salvage strategy for patients with severe peripheral arterial disease. J Vasc Surg. 2015 Sep;62(3):673-80. doi: 10.1016/j.jvs.2015.02.059. PMID 26304481